CLINICAL TRIAL: NCT00391313
Title: CuraChik : Double Blind Placebo-controlled Randomized Trial : Efficacy and Safety of Chloroquine as Therapeutic Treatment of Chikungunya Disease.
Brief Title: CuraChik : A Trial of the Efficacy and Safety of Chloroquine as Therapeutic Treatment of Chikungunya Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated Chikungunya diseases has regressed and no more patients was suffering
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006-002624-42
Record Dates: First submitted 2006-10-20; First posted 2006-10-23 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Chikungunya Virus
Keywords: Chikungunya; Chikungunya disease
MeSH Terms: conditions — Chikungunya Fever | interventions — Chloroquine

INTERVENTIONS:
Drug: Chloroquine

SUMMARY:
A severe outbreak of Chikungunya fever has been reported at La Réunion Island (France) in 2005-2006. Chikungunya is a viral disease. Chikungunya virus is an alphavirus transmitted to humans by the bite of infected mosquitoes, usually of the genus Aedes (Aedes albopictus in La Réunion).

To date, more than 266,000 cases were estimated to have occurred in the island (760,000 inhabitants). Most of cases are expressed as a mild disease, with intense fever and arthralgias, with rare but serious complications (encephalitis, liver, cardiac or renal failures.) having required a hospitalization in an intensive care unit. 273 of such serious cases (immediately life threatening condition) have been reported among the cases, in patients aged over 10 days (59% were 65+ age old). Chikungunya was proven in 246 serious cases; 101 patients had comorbidities, and 27% of confirmed cases eventually died. In addition 44 cases of mother-to-child infections were reported and 40 were confirmed (one died).

To date, in 248 death certificates, chikungunya was reported as the direct or indirect cause of death, with a median age of 79, range 0-102, and a sex-ratio (M/F) of 0.95. InVS, in collaboration with Inserm (French NIH) also reported (by June 6, 2006) a significant excess of mortality (from all causes) during the major outbreak which occurred from December, 2005 (+10%) to April, 2006 (10.1%), with a peak of excess mortality reached in February (+34.4%), concommitant to the peak of incidence.

Today, there is no antiviral treatment against Chikungunya. We showed from ex-vivo studies (in a sensitive model of cells culture to the viral infection) that chloroquine provides a significant inhibition on the replication of the Chikungunya virus. This efficacy seemed also to be reached at a plasmatic concentration of similar order of magnitude as recommended for treating malaria with this drug.

This trial aims to assess efficacy and safety of chloroquine as as therapeutic treatment of chikungunya disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of more than 18 years and less than 66 years (men and nonpregnant women, without counter-indications) voluntary to take part in of the study, residing at the Reunion Island, having a body weight equal to or higher than 60 kg for a clinical chikungunya disease diagnosed within less than 48 hours.

Exclusion Criteria:

* Pregnant Women
* More than 66 years old
* body weight less than 60 kg
* without counter-indications to chloroquine
* Renal Insufficiency
* Retinopathy
* Coeliac disease

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-05; Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier de Lamballerie, MD, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Cellule Coordination Nivachik, Saint-Pierre, Ile de La Reunion, France